CLINICAL TRIAL: NCT05759013
Title: A Randomized, Sham Controlled, Double-blinded, Multi-center Trial to Evaluate the Efficacy of the VentFree Respiratory Muscle Stimulator to Assist Ventilator Weaning in Critically Ill Patients
Brief Title: Pivotal Evaluation of Abdominal Neuromuscular Electrical Stimulation (VentFree) for Weaning From Mechanical Ventilation
Acronym: PREVENT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Liberate Medical (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LM-VF-P3; CDMRP - PR21220 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-01-16; First posted 2023-03-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-01

CONDITIONS: Respiration, Artificial; Ventilators, Mechanical
Keywords: Respiratory Muscle Stimulation; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- VentFree Respiratory Muscle Stimulator (Experimental): In the VentFree treatment group, abdominal functional electrical stimulation (FES) will be applied with a frequency of 30 hertz (Hz) and a pulse width of 350µs to cause a strong visible or palpable muscle contraction. The stimulation amplitude will be set to 90% of the participant's maximum tolerable level Discomfort associated with the maximum tolerable level will be recorded on the VAS with pain ratings from zero (no pain) to ten (worst pain). In uncommunicative patients, the maximum tolerable level will be determined as the stimulation intensity that results in a BPS >4 or CPOT >2. The stimulation amplitude will be titrated for each participant and each stimulation session. The stimulation amplitude will be evaluated every 10 (± 2) minutes after the start of each stimulation session and adjusted as necessary to maintain a consistent level of visual contraction and to ensure that the stimulation intensity remains within the participant's maximum tolerable level.
  Interventions: Device: Breath synchronized abdominal FES
- Sham Respiratory Muscle Stimulator (Sham Comparator): In the sham group, abdominal functional electrical stimulation (FES) will be set to cause sensory stimulation but no muscle contraction. Abdominal FES will be applied with a frequency of 30 hertz (Hz), a pulse width of 350 µs and a stimulation amplitude that does not cause abdominal wall muscle contraction. The stimulation amplitude will initially be set at 10 mA and reduced in steps of 2 milliamp (mA) until no muscle contraction is seen.
  Interventions: Device: Sham breath synchronized abdominal FES

INTERVENTIONS:
Device: Breath synchronized abdominal FES — Active abdominal stimulation will be applied for 30 minutes twice per day (minimum of four hours between stimulation sessions), for a minimum of five days per week, for 28 days or ICU discharge, whichever comes first.
  Other Names: VentFree Respiratory Muscle Stimulator
  Arms: VentFree Respiratory Muscle Stimulator
Device: Sham breath synchronized abdominal FES — Sham abdominal stimulation will be applied for 30 minutes twice per day (minimum of four hours between stimulation sessions), for a minimum of five days per week, for 28 days or ICU discharge, whichever comes first.
  Arms: Sham Respiratory Muscle Stimulator

SUMMARY:
The objective of this study is to evaluate the efficacy of the VentFree Respiratory Muscle Stimulator (VentFree) in critically ill adult patients who require invasive mechanical ventilation, when compared to sham.

DETAILED DESCRIPTION:
Approximately 40% of patients who receive invasive ventilation require more than four days of ventilator support. Every additional day of mechanical ventilation results in increased patient morbidity and mortality and increased economic cost. Mechanically ventilated patients often develop expiratory muscle weakness, which has been linked to failed extubation and weaning.

Neuromuscular electrical stimulation (NMES) uses electrical pulses to induce a muscle contraction and has been shown to reduce or retard muscle atrophy. NMES applied to the abdominal wall muscles has been shown to improve respiratory function and assist ventilator weaning in spinal cord injury. Liberate Medical has previously shown that NMES applied to the abdominal wall muscles in synchrony with exhalation is feasible in patients receiving invasive mechanical ventilation. This study is a pivotal evaluation of the efficacy of exhalation synchronized abdominal NMES to assist ventilator weaning in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 22 years of age.
2. Participant has been receiving invasive mechanical ventilation for ≥ 24 hours.

Exclusion Criteria:

1. Participant has been receiving invasive mechanical ventilation for > 96 hours.
2. Participant is scheduled or expected to be disconnected from mechanical ventilation ≤ 24 hours after enrollment.
3. Participant was intubated for ≥ 24 hours during a prior episode of invasive mechanical ventilation during current hospitalization.
4. Participant has a BMI ≥ 40 Kg/m2.
5. Participant has no contraction of the abdominal wall muscles in response to abdominal FES as determined by ultrasound.
6. Participant has a pre-existing neuromuscular or muscular disorder that could affect the respiratory muscles (e.g., spinal cord injury or Guillain-Barré syndrome).
7. Participant has had open abdominal surgery ≤ 4 weeks prior to enrollment.
8. Participant has open or damaged skin at area of electrode placements.
9. Participant has a pacemaker and/or implanted electronic device.
10. Participant is known or expected to be pregnant. NOTE: A negative urine or blood pregnancy test will be documented during screening for women of child-bearing potential.
11. Participant is actively pharmacologically paralyzed at the time of enrollment. NOTE: Participants receiving neuromuscular blockers may be enrolled after a ≥ 12-hour washout period.
12. Participant is tracheostomized at the time of enrollment.
13. Participant is on home non-invasive ventilation (except for CPAP or BiPAP for obstructive sleep apnea).
14. Participant is receiving or expected to receive comfort measures (palliative, hospice, comfort care, etc.) at the time of screening or enrollment.
15. Participant is participating in any of the following:

    * A study with the same or similar primary endpoint
    * A study investigating electrical stimulation or respiratory muscle therapy
    * Any study in which the investigator determines may interfere with the results of this study
16. Participant is unable or unwilling to comply with protocol requirements, including assessments, tests, and follow-up visits.
17. Participant has any other medical condition which in the opinion of the Investigator will make participation medically unsafe or interfere with the study results.
18. Participant or legally authorized representative is unwilling to provide written informed consent.
19. Participant or legally authorized representative is unable to provide written informed consent.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time from first FES treatment administration to successful liberation during the treatment period of 28 days or until ICU discharge, whichever occurs first. | From first FES treatment to 28 days or ICU discharge, whichever occurs first
  Successful liberation is defined as disconnection from mechanical ventilation that does not require invasive mechanical ventilation in the subsequent 7 days after disconnection, or until ICU discharge, or until live hospital discharge, whichever occurs first.

SECONDARY OUTCOMES:
Cough peak flow | At 24 hours post-extubation
  Cough peak flow measurement
Maximum expiratory pressure | At 24 hours post-extubation
  Maximum expiratory pressure measurement
Incidence of device-related adverse events | From date of first FES treatment administration to date of hospital discharge or 90 days after treatment, whichever occurs first
  Number of device-related adverse events
Time from first FES treatment administration to ICU discharge | From date of first FES treatment administration to date of ICU discharge or 90 days after treatment, whichever occurs first
  Duration of first FES treatment administration to ICU discharge
Time from first FES treatment administration to hospital discharge | From date of first FES treatment administration to date of hospital discharge or 90 days after treatment, whichever occurs first
  Duration of first FES treatment administration to hospital discharge
Incidence of patients who were successfully liberated from mechanical ventilation | From date of first FES treatment administration to date of hospital discharge or 90 days after treatment, whichever occurs first
  Number of of patients who were successfully liberated from mechanical ventilation
Incidence of re-intubations | From date of first FES treatment administration to 90 days after treatment
  Number of re-intubations
Incidence of readmissions to the ICU | From date of first FES treatment administration to 90 days after treatment
  Number of readmissions to the ICU
Incidence of readmissions to the hospital | From date of first FES treatment administration to 90 days after treatment
  Number of readmissions to the hospital
Incidence of acute respiratory infections | From date of first FES treatment administration to date of hospital discharge or 90 days after treatment, whichever occurs first
  Number of participants that had diagnosed acute respiratory infections
Incidence of hospital acquired infections | From date of first FES treatment administration to date of hospital discharge or 90 days after treatment, whichever occurs first
  Number of participants that had diagnosed hospital acquired infections
Incidence of tracheostomy | From date of first FES treatment administration to date of ICU discharge or 90 days after treatment, whichever occurs first
  Number of participants that underwent tracheostomies
Mortality | From Date of first FES treatment administration to date of hospital discharge or 90 days after treatment, whichever occurs first
  Number of Deaths
Maximum inspiratory pressure | At 24 hours post-extubation
  Maximum inspiratory pressure measurement
Mobility as assessed by the ICU Mobility Scale | Date of ICU discharge or 90 days after treatment, whichever occurs first
  Mobility assessment score from 0 (participant is unable to move) - 10 (participant is able to walk independently)
Quality of life as assessed by EQ-5D (Quality of Life Survey) | At 90 days after treatment
  Five (5) level Quality of Life assessment ranging from Level 1 (indicating no problem) to Level 5 (indicating unable to/extreme problems)

CONTACTS AND LOCATIONS:
Overall Officials: Angus Mclachlan, PhD, Study Director — Liberate Medical
Locations (27):
- United States (15):
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - University of Florida College of Medicine - Jacksonville, Jacksonville, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Loyola University, Maywood, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Weill Cornell Medicine / New York Presbyterian Hospital, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann, Houston, Texas
  - Providence Regional Medical Center, Everett, Washington
- Australia (5):
  - Monash Medical Centre, Clayton
  - Nepean Hospital, Kingswood
  - St. George Hospital, Kogarah
  - Prince of Wales Hospital, Randwick
  - Royal North Shore Hospital, St Leonards
- France (3):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Saint Joseph Saint Luc, Lyon
  - Pitié-Salpêtrière University Hospital, Paris
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis (JBZ), 's-Hertogenbosch
  - Canisius Wilhelmina Ziekenhuis (CWZ), Nijmegen
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No